CLINICAL TRIAL: NCT03863808
Title: Effect of Cognitive Behavioral Therapy on Chronic Low Back Pain With Sensitization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marwa Elsayed (Other)
Collaborators: MTI University (Other)
Responsible Party: Sponsor-Investigator, Marwa Elsayed, Effect of Cognitive Behavioral Therapy on Chronic Low Back Pain with sensitization., MTI University
Organization: MTI University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 118992148
Record Dates: First submitted 2018-09-23; First posted 2019-03-05 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Chronic Low Back Pain; Central Sensitisation
Keywords: Cognitive Behavioural Therapy; Flexion Relaxation Phenomenon; Electromyography; Biofeedback; Functional Training
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioural Therapy (Experimental): Following assessment a one on one session will be given comprising education cognitively targeting false ideas and beliefs on the nature of pain, differentiating nociception due to a painful stimulus and the transition of such a stimulus to a centrally sensitized experience due to misinformation, maladaptive behaviour and fear avoidance. Upon completion of the session assessment using the NPQ will be done to assess the understanding of the patient and further address any shortcomings in future exercise sessions.
  Another SEMG recording of the Flexion Relaxation phenomenon will be upon completion of the educational session and a SEMG biofeedback session will begin to help the patient regain their sense of control over their body and function.
  After the SEMG biofeedback session a graded exposure exercise program of strengthening and functional training starting from the least feared movements to the most over 10 sessions over 5 weeks.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Strengthening and Core Stability (Active Comparator): Following assessment 12 sessions over 6 weeks will start, focusing on strengthening exercises of the transversus abdominis and lumbar multifidus muscles (Angela Searle, 2015).
  Exercises will be graduated according to the patient pain tolerance.
  Interventions: Other: Strengthening exercises

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — Following assessment a one on one session will be given comprising education cognitively targeting false ideas and beliefs on the nature of pain, differentiating nociception due to a painful stimulus and the transition of such a stimulus to a centrally sensitized experience due to misinformation, maladaptive behaviour and fear avoidance. Upon completion of the session assessment using the NPQ will be done to assess the understanding of the patient and further address any shortcomings in future exercise sessions.
  Another SEMG recording of the Flexion Relaxation phenomenon will be upon completion of the educational session and a SEMG biofeedback session will begin to help the patient regain their sense of control over their body and function.
  After the SEMG biofeedback session a graded exposure exercise program of strengthening and functional training starting from the least feared movements to the most over 10 sessions over 5 weeks.
  Other Names: SEMG Biofeedback
  Arms: Cognitive Behavioural Therapy
Other: Strengthening exercises — Strengthening exercises in a gradual manner to the Multifidus and Transversus Abdominis muscles.
  Arms: Strengthening and Core Stability

SUMMARY:
PURPOSE:

The main objectives of the study are:

1. To find the efficacy of using cognitive behavioural therapy on chronic low back pain with central sensitization.
2. To assist in planning an ideal physical therapy rehabilitation program for these patients.

BACKGROUND:

Recent research has shown that CLBP is a multifactorial disorder comprising psychosocial factors like pain catastrophization, fear avoidance and central sensitization. Central sensitization has been defined as "An amplification of neural signaling within the central nervous system that elicits pain hypersensitivity", and "increased responsiveness of nociceptive neurons in the central nervous system to their normal or subthreshold afferent input".

Maladaptive behavior, false beliefs and misinformation regarding the cause of the pain are all contributing factors to the chronicity of LBP.

Central sensitization has been attributed to cortical reorganization and amplification of the somatosensory representation of the back causing increased pain and further contributing to the maladaptive behavior and beliefs.

Cognitive behavioral treatment has been an important intervention for psychological disorders for decades and recently has gained a lot of interest as an intervention for chronic pain in general and CLBP in specific.

HYPOTHESES:

It will be hypothesized that: Cognitive behavioural therapy will have a significant effect on centrally sensitized pain intensity and disability.

RESEARCH QUESTION:" Does cognitive behavioral therapy have a significant effect on chronic low back pain with central sensitization"

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18- 50.
2. Patient must have experienced low back pain for at least 3 months.
3. Patient must have a score above or equal 40 in the Central Sensitization Inventory (CSI) (Neblett R. C., 2013) (Neblett R, 2015) (Neblett H. M., 2016) (R. De Pauw, 2015) (Mayer TG N. R., 2012) .
4. Patient must have a score of 3 and above on the Numerical Pain Rating Scale.

Exclusion Criteria:

* Patients were excluded if they had taken pain medications on the day of the assessment.
* Patient who had serious spinal pathologies, such as fractures, tumors or inflammatory diseases, such as ankylosing spondylitis, narrowing of spinal canal and other conditions or severe cardiorespiratory diseases.
* Uncontrolled mental health condition that prevents successful compliance.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
The Oswestry disability index | Upto 24 weeks of treatment
  The Oswestry Disability Index (ODI) is one of the most commonly used outcome measures for individuals with low back pain (LBP) (Fairbank JC, 2000) .The ODI shows good construct validity; internal consistency is rated as acceptable; test-retest reliability and responsiveness have been shown to be high; and burden of administration is low. The ODI is a self-administered questionnaire that requires 5 minutes to complete and 1 minute to score.

SECONDARY OUTCOMES:
The fear avoidance beliefs questionnaire | Upto 24 weeks of treatment
  FABQ was developed by Waddell to investigate fear-avoidance beliefs among LBP patients in the clinical setting. This survey can help predict those that have a high pain avoidance behavior. The FABQ consists of 2 subscales, which are reflected in the division of the outcome form into 2 separate sections. The first subscale (items 1-5) is the Physical Activity subscale (FABQPA), and the second subscale (items 6-16) is the Work subscale (FABQW). Scoring the Physical Activity subscale (FABQPA) Sum items 2, 3, 4, and 5 (the score circled by the patient for these items). Scoring the Work subscale (FABQW) Sum items 6, 7, 9, 10, 11, 12, and 15.

OTHER OUTCOMES:
The numerical rating scale (NRS) | Upto 24 weeks of treatment
  The NRS evaluates levels of pain intensity using an 11-point scale (range 0-10), with 0 being classified as "no pain" and 10 "pain as bad as could be." Pain evaluation was assessed verbally by having people report pain intensity for the last 7 days as a criterion for inclusion in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- MTI University, Cairo, Mokattam, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Only consented information will be shared.

REFERENCES:
- [Result] . Airaksinen O, B. J.-M. (2006). European guidlines for the management of chronic nonspecific low back pain. Eur spine, 192-300. .: The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. . (2011). Arch Phys Med Rehabil, 2041-56. Ahern DK, F. M. (1988). Comparison of lumbar paravertebral EMG patterns in chronic low back pain patients and non-patient controls. Pain, 153-160. Airaksinen O, B. J.-M. (2006). European guidlines for the management of chronic nonspecific low back pain. Eur spine, 192-300. Angela Searle, M. S. (2015). Exercise interventions for the treatment of chronic low back pain: A systematic review and meta-analysis of randomised controlled trials. Clinical Rehabilitation, 1-13. Balagué F, M. A. (2012). Non specific low back pain. lance, 482-491. Clarke CL, R. C. (2011). Pain neurophysiology education for the management of individuals with chronic low back pain: systematic review and meta-analysis. Manual Therapy, 544-549. Cohen JE, G. V. (1994). Group education interventions for people with low back pain. An overview of the literature. Spine , 1214-22. Dagenais S, C. J. (2008). A systematic review of low back pain cost of illness studies in the United States and internationally. Spine, 8-20. DC, M. V. (2008). Psychometric properties and clinical usefulness of the Oswestry Disability Index. Journal of Chiropractice medicine, 161-163. Delitto. (2005). Research in low back pain: Time to stop seeking the elusive